CLINICAL TRIAL: NCT03610776
Title: Role of Visual Cues in the Regulation of Portion Size and the Cephalic Satiety Response in Lean and Overweight Subjects
Brief Title: Effect of Tableware Visual Cues on Portion Control and Eating Rate
Acronym: PORTIONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Gobierno de Navarra (Unknown); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Precise Portions Nutrition Learning Systems (Unknown); University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CIN-01-17
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-10

CONDITIONS: Portion Size
Keywords: Portion control plate; Visual attention; Eating rate; Cephalic satiety response

STUDY DESIGN:
Intervention Model Description: Randomised, cross-over (within-subjects) design.
Masking Description: Masking is not possible due to the nature of the intervention (portion control vs. conventional plate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portion control plate (Experimental): Portion control plate first (50% of subjects experiment with this plate first)
  Interventions: Device: Portion control plate
- Conventional plate (Active Comparator): Conventional plate first (50% of subjects experiment with this plate first)
  Interventions: Device: Conventional plate

INTERVENTIONS:
Device: Portion control plate — Portion control plate including demarcations and pictures for recommended amounts of main food groups (starch, protein and vegetables), 25 cm in diameter, enamel, white background.
  Other Names: Calibrated plate
  Arms: Portion control plate
Device: Conventional plate — Conventional plate without demarcations or images, 25 cm in diameter, enamel, white.
  Other Names: Control plate
  Arms: Conventional plate

SUMMARY:
Randomised within subjects cross-over study (n=94) exploring the cognitive and physiological processes associated with portion control. Participants will eat a self-served lunch using a portion control plate vs. a conventional (control) plate on two separate occasions under a controlled laboratory environment. Portion size, meal micro-structure, attention, memory and satiety markers will be analysed. The portion control plate is a prototype designed in collaboration with the commercial partner for this study and is based on published evidence. It includes sectors and pictures indicating amounts to serve from starchy food, protein and vegetables. The control plate will be of the same background colour, size and shape but without any pictures or demarcations. The main study outcome is attention time on areas of interest in the plate corresponding to main foods groups, across plate conditions.

DETAILED DESCRIPTION:
The size and design of tableware have been proposed as a potentially effective strategy to modulate how much is eaten at a meal. The mechanisms by which specific tableware may work however are not known, in particular the cognitive processes associated with visual stimuli. In this covert trial, 68 women (34 overweight or obese) and 26 lean men (exploratory sub-study) will self-serve and consume food from a laboratory buffet using a portion control plate with visual stimuli for appropriate amounts of main food groups, or a conventional plate, on two different days in random order. On both sessions participants will complete behavioural and cognitive tests to measure visual attention during the meal (eyetracking device), meal microstructure (Universal Eating Monitor), episodic memory for portion sizes (computerised test), portion size choice, food intake, subjective appetite and satiety, cephalic and intestinal satiety responses. Further behavioural tests include meal liking, expected satiety, portion size perceptions and tool acceptance ratings. The main study outcome is difference in proportional dwell time on areas of interest in the plate corresponding to main foods groups (women), or difference in bite size (men) across conditions. Secondary outcomes for all subjects include: portion size for overall meal and meal components, eating rate, bite size, deceleration rate, portion size memory error, portion size norms, portion control self-efficacy, tool acceptance, energy compensation for the rest of the day, plus blood insulin, glucose, pancreatic polypeptide and ghrelin up to 90 min post-meal (sub-sample of 34 women, 50% being overweight/obese). Analyses by gender and BMI sub-groups will be applied when possible. The results of this study will help to better understand the potential mechanisms by which portion control tools with visual cues may work, and to improve the design of current instruments for their application in nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 18-60 years.
2. For women, having a BMI between 18.5 and 35 kg/m2 (both included); for men having a BMI between 18.5 and 25 kg/m2 (both included).
3. Healthy as determined from the self-reported medical history or when a clinical condition exists, when this is considered to be irrelevant for the study by the study medical doctor.
4. Not taking any medication that may affect sight, gastro-intestinal function or appetite. Volunteers taking medication for clinical conditions that may affect the above functions will be eligible if they report no side effects and the dose has been stable for at least 3 months prior to commencement of the study.
5. Consuming breakfast and lunch regularly (at least 5 days per week).
6. Liking of the study foods defined by a score of >40 mm of the Liking VAS questionnaire, for each compulsory meal component.
7. Able to consume food without the need for prescription glasses (contact lenses are allowed).
8. Able to understand and be willing to sign the informed consent form and to follow all the study procedures and requirements.

Exclusion Criteria:

1. Deficient nutrition or hydration status at the time of recruitment.
2. Abnormal gastro-intestinal function or structure such as malformation, angiodysplasia, active peptic ulcer, and chronic inflammatory or malabsorptive diseases, even if at the time of recruitment the volunteer is not taking medication for such conditions (e.g. anti-inflammatory drugs).
3. History of gastro-intestinal surgery with permanent sequels (i.e. gastroduodenostomy).
4. History of liver disease.
5. History of cancer or receiving treatment for cancer.
6. Diabetes mellitus.
7. Food allergy, food restriction or avoidance of any of the study foods (e.g. vegetarian).
8. History of mental illness, or being under active treatment for mental illness (e.g. psychiatric disorder), whenever their condition affects their ability to comprehend or follow the requirements of the study in full, or when their condition affects short-term memory (e.g. Alzheimer disease).
9. Presence of an eating disorder defined as a score >19 on the Eating Attitudes Test (EAT-26).
10. Diagnosed or suspected epilepsy or photosensitive epilepsy (e.g. experiencing an "aura" or odd sensations while watching images or patterns on a computer screen).
11. Wearing a pacemaker or other medical electronic device.
12. Currently dieting to lose weight.
13. Smoking > 7 cigarettes per week.
14. Consuming >14 units of alcohol intake per week in women, or >21 units per week in men.
15. Performing >9 h of intense physical activity per week.
16. Pregnancy or lactation.
17. Having received formal portion size education as part of a university degree (e.g. Dietetics, Human Nutrition, Psychology if relevant).
18. Being familiar with the nature of the covert measures involved in the study (i.e. measure of eating speed and bite size).
19. Volunteers for which insufficient collaboration may be foreseen, or whom the investigator has grounds to believe that they may experience difficulty in following the study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Dwell time difference (women) | Month 24
  Difference in proportional dwell time on three areas of interest in the plate corresponding to main food groups i.e. starch, protein and vegetables, measured in milliseconds, as a proxy for attention levels, between the Portion Control Plate condition and the conventional plate condition.
Bite size difference (men) | Month 24
  Difference in the amount of food loaded on the fork estimated from the difference in grams between two consecutive weight records as measured by the Universal Eating Monitor, between the Portion Control Plate condition and the conventional plate condition.

SECONDARY OUTCOMES:
Eating rate difference | Month 24
  Difference in grams of food consumed per minute as measured by the Universal Eating Monitor, between conditions (Portion Control Plate vs. conventional plate).
Bite size difference (women) | Month 24
  Difference in the amount of food loaded on the fork estimated from the difference in grams between two consecutive weight records as measured by the Universal Eating Monitor, between conditions (Portion Control Plate vs. conventional plate).
Deceleration rate difference | Month 24
  Difference in the change in eating rate over the course of the meal measured in grams per squared second, as recorded by the Universal Eating Monitor, between conditions (Portion Control Plate vs. conventional plate).
Meal duration difference | Month 24
  Difference in the duration of the meal in minutes, starting when the investigator places the food on the table and finishing when the volunteer pressed the bell, between conditions (Portion Control Plate vs. conventional plate).
Dwell time difference (men) | Month 24
  Difference in proportional dwell time on three areas of interest in the plate corresponding to main food groups i.e. starch, protein and vegetables, measured in milliseconds, as a proxy for attention levels, between conditions (Portion Control Plate vs. conventional plate).
Difference in portion size at meal | Month 24
  Difference in portion sizes in grams for the complete meal and for each meal component (i.e. rice, vegetables, meatballs, bread, fruit, condiments and water), between conditions (Portion Control Plate vs. conventional plate).
Percent memory reconstruction error (Portion Control Plate) | Month 21
  Percent error between recalled and real portion size calculated by subtracting the recalled portion size for each meal component at 3 hours post-meal, from the actual portion sizes chosen during the test meal and dividing by the actual portion size, using data from a computer-based memory reconstruction task (XnConvert software), for the Portion Control Plate condition. Interpreted as 0% = perfect match between recalled and actual portion size.
Percent memory reconstruction error (conventional plate) | Month 21
  Percent error between recalled and real portion size calculated by subtracting the recalled portion size for each meal component at 3 hours post-meal, from the actual portion sizes chosen during the test meal and dividing by the actual portion size, using data from a computer-based memory reconstruction task (XnConvert software), for the conventional plate condition. Interpreted as 0% = perfect match between recalled and actual portion size.
Percent memory reconstruction error difference | Month 24
  Difference in the percent memory reconstruction error for each meal component at 3 hours post-meal, between the Portion Control Plate and the conventional plate condition.
Percent energy compensation (EC) | Month 21
  Energy adjustment after the meal and for the remaining of the day, calculated from food intake data collected via an 8h food diary and using a published algorithm (Almiron-Roig et al. 2013). Interpreted as EC of 100% = perfect compensation; <100% = undercompensation; >100% overcompensation.
Percent energy compensation difference | Month 24
  Difference in percent energy compensation after the meal and for the remaining of the day, between conditions (Portion Control Plate vs. conventional plate).
Portion size norms | Month 21
  Visual analogue scale ratings (0 -100 mm) for habitual portion size for the meal, rice, vegetables and meatballs consumed during the test meal. Interpreted as: a score of 50 mm = the chosen portion equals the habitual portion size; >50 mm = chosen portion is smaller than habitual; <50 mm = chosen portion is larger than habitual.
Portion size norms difference | Month 24
  Difference in Visual Analogue Scale ratings for portion size norms for the whole meal, rice, vegetables and meatballs between conditions (Portion Control Plate vs. conventional plate).
Liking for the meal differences | Month 24
  Difference in visual analogue scale ratings (0-100 mm) for Liking of the meal after consumption between conditions (Portion Control Plate vs. conventional plate).
Baseline subjective appetite | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived hunger before the meal (time 0)
Baseline subjective satiety | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived fullness before the meal (time 0)
Baseline subjective thirst | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived thirst before the meal (time 0)
Baseline subjective nausea | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived nausea before the meal (time 0)
Post-meal subjective appetite | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived hunger immediately after the meal (time 1)
Post-meal subjective satiety | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived fullness immediately after the meal (time 1)
Post-meal subjective thirst | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived thirst immediately after the meal (time 1)
Post-meal subjective nausea | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived nausea immediately after the meal (time 1)
3 h subjective appetite | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived hunger 3 hours after consuming the meal (time 2)
3 h subjective satiety | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived fullness 3 hours after consuming the meal (time 2)
3 h subjective thirst | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived thirst 3 hours after consuming the meal (time 2)
3 h subjective nausea | Month 21
  Visual analogue scale ratings (0-100 mm) for perceived nausea 3 hours after consuming the meal (time 2)
Difference in subjective appetite and satiety scores | Month 24
  Difference in scores of visual analogue scale ratings (0-100 mm) for perceived hunger, fullness, thirst and nausea at baseline, post-meal and 3 hours after consuming the meal, between conditions (Portion Control Plate vs. conventional plate).
Difference in expected satiation for the meal | Month 24
  Difference in visual analogue scale rating (0-100 mm) before consuming the meal, between conditions (Portion Control Plate vs. conventional plate).
Baseline blood glucose | Month 21
  Blood glucose levels before starting the meal
Post-meal blood glucose | Month 21
  Blood glucose levels at 5, 10, 30, 60 and 90 min after starting the meal
Difference in post-meal blood glucose | Month 21
  Difference in blood glucose levels at 5, 10, 30, 60 and 90 min after starting the meal between conditions (Portion Control Plate vs. conventional plate).
Baseline blood insulin | Month 21
  Blood insulin levels before starting the meal
Post-meal blood insulin | Month 21
  Blood insulin levels at 5, 10, 30, 60 and 90 min after starting the meal
Difference in post-meal blood insulin | Month 24
  Difference in blood insulin levels at 5, 10, 30, 60 and 90 min after starting the meal between conditions (Portion Control Plate vs. conventional plate).
Baseline blood pancreatic polypeptide | Month 21
  Blood pancreatic polypeptide levels before starting the meal
Post-meal blood pancreatic polypeptide | Month 21
  Blood pancreatic polypeptide levels at 5, 10, 30, 60 and 90 min after starting the meal
Difference in post-meal blood pancreatic polypeptide | Month 24
  Difference in blood pancreatic polypeptide levels at 5, 10, 30, 60 and 90 min after starting the meal between conditions (Portion Control Plate vs. conventional plate).
Baseline blood ghrelin | Month 21
  Blood ghrelin levels before starting the meal
Post-meal blood ghrelin | Month 21
  Blood ghrelin levels at 5, 10, 30, 60 and 90 min after starting the meal
Difference in post-meal blood ghrelin | Month 24
  Difference in blood ghrelin levels at 5, 10, 30, 60 and 90 min after starting the meal between conditions (Portion Control Plate vs. conventional plate).
Body Mass Index | Month 18
  Weight in kilograms divided by height in squared meters measured at the start of the trial.
Age | Month 18
  Age in years measured at the start of the trial.
Eating behaviour profile from the Three Factor Eating Questionnaire (TFEQ) | Month 21
  Restraint, disinhibition and susceptibility to hunger scores from the Three Factor Eating Questionnaire for the Spanish population (Sánchez-Carracedo et al. 1999, Psicol Conduct 7:393-416) measured at the end of the trial.
Eating behaviour profile from the Eating Attitudes Test (EAT-26) | Month 18
  Susceptibility to eating disorders score using the Eating Attitudes Test (EAT-26) the Spanish population (Rivas et al. 2010; Span J Psychol 13:1044-1056) measured at the start of the trial.
Difference in portion control self-efficacy | Month 24
  Difference in portion control self-efficacy score derived from the Portion Control Self-Efficacy Scale (Fast et al.2015) between conditions (Portion Control Plate vs. conventional plate). The scale ranges from 1 to 5. A combined score will be obtained for questions 1,2, 3, 5, 7,8 and the reverse of questions 4 and 6, by adding up all the scores from each of the 8 Likert scales, and dividing the sum by 8. A score between 1-2.5 will be interpreted as 'none to low self-efficacy'; a score between 2.5-3.5 will be interpreted as 'neutral self-efficacy', a score between 3.5-5 will be interpreted as 'medium to high self-efficacy'.
Difference in portion tool acceptance | Month 24
  Difference in portion tool acceptance score derived from a published questionnaire (Almiron-Roig et al., 2016) between conditions (Portion Control Plate vs. conventional plate). A combined score will be obtained for questions a, b, c, e, f, g and the reverse of d by adding up all the scores from each of the 4 Likert scales, and dividing the sum by 7. A score between 1-2.5 will be interpreted as 'none to low acceptance'; a score between 2.5-3.5 will be interpreted as 'neutral acceptance', a score between 3.5-5 will be interpreted as 'medium to high acceptance'.
Self-reported ethnicity | Month 18
  Ethnicity group defined using a check-list, measured at the start of the trial.
Household composition | Month 18
  Number of adults and children aged 18 or less living in the same household (checklist) measured at the start of the trial.
Take away food consumption | Month 18
  Frequency of take away food consumption (checklist), measured at the start of the trial.
Home-made meal consumption | Month 18
  Frequency of home-made meal consumption (checklist), measured at the start of the trial.
Cooking pattern | Month 18
  Cooking for self only vs. cooking for self and others (checklist), measured at the start of the trial.
Previous experience with portion tools | Month 18
  Previous experience with portioning utensils, portion control tools, measuring utensils etc. (open ended question), measured at the start of the trial.
Food intake for remaining of the day | Month 21
  8h food record to complete after the laboratory test meal, for both conditions (Portion Control Plate and conventional plate).

OTHER OUTCOMES:
Meal component palatability scores | Month 18
  Visual analogue scale ratings (0-100 mm) for liking of the rice, peas, carrots and meatballs, measured during a sensory test at the start of the trial (laboratory screening session).
Smoking frequency | Month 18
  Self-reported number of cigarettes per day measured at the start of the trial (telephone screening interview).
Physical activity frequency | Month 18
  Self-reported number of hours of moderate to intense physical activity per week, measured at the start of the trial (telephone screening interview).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Almiron-Roig, PhD, Principal Investigator — University of Navarra
Locations (1):
- Centre for Nutrition Research, University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Almiron-Roig E, Dominguez A, Vaughan D, Solis-Trapala I, Jebb SA. Acceptability and potential effectiveness of commercial portion control tools amongst people with obesity. Br J Nutr. 2016 Dec;116(11):1974-1983. doi: 10.1017/S0007114516004104. Epub 2016 Dec 15. PMID 27976604
- [Background] Almiron-Roig E, Palla L, Guest K, Ricchiuti C, Vint N, Jebb SA, Drewnowski A. Factors that determine energy compensation: a systematic review of preload studies. Nutr Rev. 2013 Jul;71(7):458-73. doi: 10.1111/nure.12048. Epub 2013 Jun 10. PMID 23815144
- [Background] Fast LC, Harman JJ, Maertens JA, Burnette JL, Dreith F. Creating a measure of portion control self-efficacy. Eat Behav. 2015 Jan;16:23-30. doi: 10.1016/j.eatbeh.2014.10.009. Epub 2014 Nov 1. PMID 25464062
- [Derived] Vargas-Alvarez MA, Al-Sehaim H, Brunstrom JM, Castelnuovo G, Navas-Carretero S, Martinez JA, Almiron-Roig E. Development and validation of a new methodological platform to measure behavioral, cognitive, and physiological responses to food interventions in real time. Behav Res Methods. 2022 Dec;54(6):2777-2801. doi: 10.3758/s13428-021-01745-9. Epub 2022 Jan 31. PMID 35102518